CLINICAL TRIAL: NCT00979485
Title: Microparticles in Pediatric Inflammatory Bowel Disease
Brief Title: Microparticles in Pediatric Inflammatory Disease
Status: Terminated | Type: Observational
Why Stopped: initial results suggest no significant trends will be observed with completion of study
Sponsor: Indiana University (Other)
Responsible Party: Steven Steiner, MD, Indiana University
Other Study IDs: 0906-75
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Pediatric IBD; Microparticles
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to provide data correlating levels of microparticles that circulate in the blood and disease activity in children with inflammatory bowel disease (IBD). The hypothesis is that circulating microparticles will be higher in children with active IBD, show inflammatory activity, and will be low in patients in remission as well as in healthy controls.

DETAILED DESCRIPTION:
Once the response of microparticles to inflammation is defined in this patient population, the microparticles can be used as biomarkers of disease activity and could potentially use microparticles as targets of therapeutic agents.

This cross sectional study will enroll 15 Crohn's patients (5 inactive, 5 mild, 5 moderate-severe disease based on the pediatric Crohn's disease activity index), 15 Ulcerative Colitis patients (5 inactive, 5 mild, 5 moderate-severe disease based on the pediatric ulcerative colitis activity index), and 10 healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Children with IBD based on endoscopic, histologic, radiologic, or laboratory data
* Ages between 8 and 17 years old

Exclusion Criteria:

* Anyone with a concurrent illness since infection can affect microparticle levels

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric GI clinic at Riley Hospital Pediatric well child clinic at Riley Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven ' Steiner, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana Unversity, Riley Hospital for Children, Indianapolis, Indiana, United States